CLINICAL TRIAL: NCT04405661
Title: Correlation Between Specific Gene Mutationand Local Immune Microenvironment and Immunotherapy Efficacy in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: GeneCast Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhou Chengzhi, PHD,Chief Physician, Guangzhou Institute of Respiratory Disease
Other Study IDs: NSCLC-202005
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: NSCLC
Keywords: PD-L1; NSCLC; Biomarker; mIHC; immune microenvironment; mutation; sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE tissue and whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immunotherapy for PD-L1 positive patients is still ineffective in some patients，which may be related to the complex immune microenvironment.In view of this bottleneck, further refinement of immunotyping and in-depth study of drug resistance mechanism are the most important tasks. In this observational study, we evaluated the difference of gene mutation and immune microenvironment and therapeutic effect in primary NSCLC.

DETAILED DESCRIPTION:
There are still some patients with PD-L1 positive who are ineffective in immunotherapy, which may be related to the complex immune microenvironment. In view of this bottleneck, further refinement of immunotyping and in-depth study of drug resistance mechanism are the most important tasks.

Recently, studies have shown that the core elements of tumor microenvironment that have a significant impact on immunotherapy are:1. Infiltration abundance of specific killer T cells; 2. PD-L1 expression dependent on IFN - γ pathway, down-regulation of various active molecules and up-regulation of inhibitory molecules; 3. Activation and clearance of various inhibitory T cells.

Although the classification has achieved further refinement of immune cells and molecular level, there are still some problems to be solved urgently: first, the classification of TIL cells needs further refinement, and different types of TIL infiltration have different guiding significance for prognosis; second, the subjective second-order semi quantitative scoring is often used for til count scoring, with low repeatability and different centers It is not easy for different pathologists to reach an agreement on the results of reading and interpretation. Thirdly, conventional methods are difficult to meet the requirements of tumor microenvironment analysis. In conclusion, it is urgent to develop a multi molecular marker landscape analysis system for tumor microenvironment, and establish a standardized detection process for each molecule to meet the needs of clinical positioning, quantitative and qualitative analysis for key molecular markers of immune microenvironment.

In this observational study, we evaluated the difference of gene mutation and immune microenvironment and therapeutic effect in primary NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer was diagnosed by cytology or histopathology;
* Patients to be treated with PD-1 / PD-L1 inhibitors;
* Who signed the informed consent for participating in the research plan

Exclusion Criteria:

* History of other malignancies
* Cancer meningitis in subjects
* Incomplete clinical follow-up data
* Failure to sign informed consent to participate in the research program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between specific gene mutation and immune microenvironment | up to 1year
  Correlation between specific gene mutation and immune microenvironment
Correlation between specific gene mutations and ORR and PFS in immunotherapy patients with lung cancerof lung cancer patients with immunotherapy | up to 1year
  Correlation between specific gene mutations and ORR and PFS in immunotherapy patients with lung cancer
Correlation between immune microenvironment and ORR and PFS in immunotherapy lung cancer patients | up to 1year
  Correlation between immune microenvironment and ORR and PFS in immunotherapy lung cancer patients

SECONDARY OUTCOMES:
Correlation of OS with specific gene mutation in immunotherapy of lung cancer | up to 1year
  Correlation of OS with specific gene mutation in immunotherapy of lung cancer
Correlation between immune microenvironment and OS in immunotherapy lung cancer patients | up to 1year
  Correlation between immune microenvironment and OS in immunotherapy lung cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China